CLINICAL TRIAL: NCT06007001
Title: Telerehabilitation and Tele-psychological Support in Cancer Patients: the Pilots Projects of eCAN JA
Brief Title: Telerehabilitation and Tele-psychological Support in Cancer Patients eCAN JA
Acronym: eCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sciensano (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eCAN pilots
Record Dates: First submitted 2023-06-23; First posted 2023-08-23 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Cancer; telemedicine; teleconsultation; telemonitoring; PROM; PREM
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Patients in the intervention group will receive weekly teleconsultation of 30 minutes during 8 weeks through the secure Edumeet platform. In pilot 1, tele-rehabilitation training will be performed by a remote physiotherapist and will consist of a series of rehabilitation exercises. In pilot 2, tele-psychological support will be performed by a remote psychologist and will consist of techniques for managing emotions and stress. In the intervention group, patients will also have the possibility to wear a smartwatch to automatically collect physical parameters.
  Interventions: Device: Telemedicine
- Usual care (No Intervention): Patients in the control group will receive usual care.

INTERVENTIONS:
Device: Telemedicine — Pilot 1a/b : the tele-rehabilitation intervention in BC or H&N operated patients will consist of a series of exercises. The physiotherapist during teleconsultation rehabilitation program will explain to the patient how to perform the movements and regulate breathing. Practical advice on correct and incorrect habits will also be dispensed by the physiotherapist during the teleconsultation.
  Pilot 2: the tele-rehabilitation intervention will consist of tele psychological support performed by a trained psychologist in each participating center It will consist of the learning of techniques for managing negative emotions, for relaxation and for implementing effective behavioural and coping strategies.
  For each group, the TC will be scheduled every week for 8 weeks. The session will be available on a secure platform (Edumeet). Moreover, if they agree to, patients will also wear a smart watch to monitor physical parameters such as physical activity, sleeping and heart rate.
  Arms: Telemedicine

SUMMARY:
The integration of teleconsultation (TC) and telemonitoring (TM) in cancer patients care may allow to improve person-centered care and patients' empowerment.

The eCAN JA explores the role of telemedicine tools (i.e. TC & TM) in clinical trials focusing on tele-rehabilitation and tele-psychological support in different populations of cancer patients in 10 European countries. The pilots will be conducted among 354 patients affected by breast (BC, pilot 1a), head & neck (H&N, pilot 1b) and advanced (pilot 2) cancers.

The main aim is to assess the effect of TC and TM program focused on rehabilitation and psychological support for cancer patients on patient reported outcomes measures (PROMs) in three pilots compare to usual care.

Patients will be randomly assigned either to the intervention or control groups using a 1:1 ratio. Patients in the intervention group will receive weekly TC of 30 minutes during 8 weeks through the secure Edumeet platform. In pilot 1, tele-rehabilitation training will be performed by a remote physiotherapist and will consist of a series of rehabilitation exercises. In pilot 2, tele-psychological support will be performed by a remote psychologist and will consist of techniques for managing emotions and stress. In the intervention group, patients will also have the possibility to wear a smartwatch to automatically collect physical parameters. Patients in the control group will receive usual care.

PROMs (i.e. quality of life, distress and pain) and physical parameters (i.e. physical activity, sleep quality and heart rate) will be monitored by a dedicated telemonitoring systems. A secure web platform will provide dashboard to clinicians for decision support. Patients' experience and costs data will be also collected. The results of the eCAN project will improve our knowledge on benefits and risks for TC and TM in cancer patients care.

ELIGIBILITY:
Inclusion Criteria:

* Pilot 1a: All consenting adult women, aged between 45 and 65 years old, who undergo a unilateral mastectomy plus axillary dissection for newly diagnosed breast cancer in a cancer center of participating European countries will be eligible for this study.
* Pilot 1b: All consenting adult patients, aged between 18 and 75 years old, with histopathologically proven H&N cancer who are prescheduled for an en bloc resection of the primary tumor, neck dissection, or reconstruction in a cancer center of participating European countries will be eligible for this study.
* Pilot 2: All consenting adult patients, aged between 18 and 75 years old, affected by advanced/recurrent cancer (including lung, prostate, colorectum, breast cancer, gastric, genito-urinary) will be eligible for this study.

Exclusion Criteria:

* For both study pilot 1a & 1b: Patients are ineligible to participate if they meet one of the following criteria: (I) having breast reconstruction, (II) having blindness or severe visual impairment, (III) having life expectancy of less than 3 months, (IV) having previous upper limb injury or conditions that limit upper limb range of motion (shoulder flexion (< 150°) or elbow extension/flexion (< 0/145°) respectively), (V) unable to be assigned to tele-rehabilitation due to clinical conditions requiring in-person rehabilitation, (VI) unable to sign informed consent, (VII) not having access to an internet connection, (VIII) not having access to an android smartphone or (IX) already involved in other telemedicine services. For pilot 1b, H&N cancer patients needing post-surgery radiotherapy will be excluded.
* For pilot 2: Patients are ineligible to participate if they meet one of the following criteria: (I) unable to sign informed consent; (II) present relevant cognitive deterioration; (III) performance status > ECOG 2; (IV) previous diagnosis of major depression, the presence of mood disorders will be assessed with Personal Health Questionnaire Depression Scale (PHQ-8) (13); (V) starting antidepressant pharmacological treatment in the last 4 weeks before the enrollment; (VI) taking antipsychotic treatment, (VII) not having access to an internet connection (VIII) not having access to an android smartphone or (IX) already involved in other telemedicine services.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Health related quality of life measure to 8 weeks | Every 2 weeks: week 0, 2, 4, 6, 8
  EORTC QLQ-C30 questionnaire

SECONDARY OUTCOMES:
Change from baseline Pain level to 8 weeks (for pilot 1) | weekly: week 0, 1, 2, 3, 4, 5, 6, 7, 8
  Visual Analogical Scale (VAS). The ends are defined as the extreme limits of the parameter to be measured (orientated from the left (0 the worst) to the right (100 the best).
Change from baseline Distress level to 8 weeks (for pilot 2) | weekly: week 0, 1, 2, 3, 4, 5, 6, 7, 8
  NCCN Distress thermometer.Distress is an unpleasant experience of a mental, physical, social, or spiritual nature. It can affect the way you think, feel, or act. Distress may make it harder to cope with having cancer, its symptoms, or its treatment. Please circle the number (0-10) that best describes how much distress you have been experiencing in the past week, including today.

OTHER OUTCOMES:
Change from baseline Physical activity to 8 weeks | every day, up to 8 weeks
  physical activity, number of steps, will be collected via wearable devices
Change from baseline sleep quality to 8 weeks | every day, up to 8 weeks
  The average sleep quality (light sleep, deep sleep, REM sleep) will be collected via wearable device (Garmin watche)
Change from baseline heart rate to 8 weeks | every day, up to 8 weeks
  Daily heart rate (beats per minute) trend will be collected via wearable device (Garmin watche)
Patient-reported cost | at week 9
  Costs that arose for patients will be collected using a patient-reported cost questionnaire.
PREMS - mHealth App Usability | at week 9
  usability of the teleconsultation program and telemonitoring with mHealth App Usability Questionnaire (MAUQ) for Standalone mHealth Apps Used by Patients
PREMS - telehealth usability | at week 9
  usability of the teleconsultation program and telemonitoring with TELEHEALTH USABILITY QUESTIONNAIRE (TUQ)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pace, Dr, Principal Investigator — Neuro-Oncology Unit, Regina Elena Cancer Institute, Italy
Locations (18):
- The Antwerp University Hospital (UZA), Antwerp, Belgium
- Cyprus (3):
  - German Oncology Center (GOC), Ágios Athanásios
  - CUT, Limassol
  - The Bank of Cyprus Oncology Center (BOCOC), Stróvolos
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- National Institute of Oncology, Budapest, Hungary
- Dr Steevens Hospital, Dublin, Ireland
- Italy (2):
  - The National Cancer Institute of Naples (INT Pascale), Naples
  - The Regina Elena National Cancer Institute (IFO-IRE), Roma
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauna Klinikos (KK), Kaunas
  - National Cancer Institute (NCI), Vilnius
  - Vilnius University Hospital Santaros Klinikos VULSK, Vilnius
- Portugal (3):
  - Portuguese Institute of Cancer of Coimbra (IPO), Coimbra
  - Portuguese Institute of Cancer of Lisbon (IPO), Lisbon
  - Portuguese Institute of Cancer of Porto (IPO), Porto
- The institute of Oncology Ljubljana (OIL), Ljubljana, Slovenia
- Spain (2):
  - IDIVAL, Santander
  - Andalusian Health Service, Seville

IPD SHARING:
Plan to Share IPD: No